CLINICAL TRIAL: NCT01094886
Title: A Open-Label Study of the Transition to Rivaroxaban From Low-Molecular Weight Heparin for Venous Thromboembolism Prophylaxis After Total Joint Replacement: The Safe Simple Transitions Study
Brief Title: Switching Drug Therapy for the Prevention of Blood Clot Formation From Enoxaparin to Rivaroxaban After Orthopedic Surgery for Either Total Hip or Total Knee Replacement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CR016531; RIVAROXCPK3001 (Other: Ortho-McNeil Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2010-03-25; First posted 2010-03-29 (Estimated); Results first posted 2012-02-27 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-02

CONDITIONS: Arthritis; Osteoarthritis, Knee; Osteoarthritis, Hip; Thromboembolism
Keywords: Total Hip Replacement; Total Knee Replacement; Hip Implant; Knee Implant; Joint Prosthesis; Orthopedic Surgery; Rivaroxaban; Xarelto; Blood Clot
MeSH Terms: conditions — Arthritis; Osteoarthritis, Knee; Osteoarthritis, Hip; Thromboembolism; Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 001 (Experimental): Rivaroxaban 10mg tablet daily receiving the first dose within two days after admission to the subacute unit. The total duration of combined venous blood clot prevention therapy with enoxaparin and rivaroxaban may not exceed 35 days for patients with total hip replacement or 14 days with total knee replacement
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban — 10mg tablet daily, receiving the first dose within two days after admission to the subacute unit. The total duration of combined venous blood clot prevention therapy with enoxaparin and rivaroxaban may not exceed 35 days for patients with total hip replacement or 14 days with total knee replacement

SUMMARY:
The study will describe the short-term effects the study drug, rivaroxaban, has on the body when a patient is switched from enoxaparin injection (by needle) to oral rivaroxaban (by mouth) for the prevention of blood clotting in the veins after elective total hip or total knee replacement surgery. After providing written informed consent, screening procedures will be completed to assess eligibility. After enrollment, all patients will be switched from enoxaparin to rivaroxaban. Blood samples for the short-term effects of rivaroxaban will be taken at various times while in the subacute unit. At the time of discharge, if the study doctor feels it is appropriate, an adequate supply of rivaroxaban will be provided to complete the full course of therapy. Upon completion of rivaroxaban therapy, all patients will be required to have final study procedures performed. Safety evaluations at the final visit will include clinical blood laboratory tests, a physical examination, urine pregnancy test (if applicable), recording of any adverse events including details regarding any bleeding episodes or blood clot events, and assessment of the surgical wound. All patients will return any unused study medication and study participation will be complete.

DETAILED DESCRIPTION:
The study medication, rivaroxaban, is an oral (by mouth) medication. Rivaroxaban directly inhibits one of the clotting mechanisms in the blood that is involved in the formation of blood clots in the veins in the body. The ability to inhibit blood clotting will be measured. Rivaroxaban is currently approved in the European Union by the European Medicines Agency (EMEA) for the prevention of blood clots in veins in orthopedic (bone) surgical patients who have had elective total joint (hip or knee) replacement. It is currently under review by the Food and Drug Administration (FDA) in the United States for this same indication. Enoxaparin is a medication that is injected into the fat tissue under the skin and is approved by the FDA for the treatment and prevention of blood clot formation in the veins. The goal of the study is to describe the short-term effects that the study drug has on the body when a patient is switched from enoxaparin to rivaroxaban. The study hypothesis, or theory, is that when switched from enoxaparin to rivaroxaban the ability of the body to inhibit blood clotting activity will continue. This is an open-label study which means that all persons involved in the study will know what study drug is being given to them. It is a single-arm study which means that all patients will be administered the same study medication, rivaroxaban. The study will be conducted at large orthopedic centers in the United States. All patients will have had elective total hip or total knee replacement surgery. While in the hospital, eligible patients will have been receiving enoxaparin either 30 mg twice a day or 40 mg once daily. Upon discharge from the hospital all eligible patients will require a stay in a subacute unit and continuing medication for blood clot prevention. After providing written informed consent, patients will have screening procedures completed to determine eligibility. Safety evaluations at the screening procedure will include a physical examination, vital signs, and clinical blood laboratory tests. Women, who are able to bear children, will also have a screening blood pregnancy test performed. A negative pregnancy test is needed to be in the study. Just before receiving the first dose of rivaroxaban, 10 mg, blood sampling for the short-term effects of rivaroxaban will begin and continue at various times. All patients will receive 10 mg of rivaroxaban daily. In addition, the study doctor will do an assessment of the surgical wound. At the time of discharge from the subacute unit, if the study doctor feels it is appropriate, an adequate supply of rivaroxaban will be provided to complete the full course of therapy. If a patient withdraws his/her consent prior to completion of the study, the appropriate course of blood clot prevention therapy will be prescribed by the study doctor. Upon completion of rivaroxaban therapy, all patients will be required to have final study procedures performed. Those patients who continue oral rivaroxaban after discharge from the subacute unit will be required to return for an office visit for final study procedures either at the time of completion of rivaroxaban therapy or at the surgical follow-up visit. Patients who have rivaroxaban discontinued prior to discharge from the subacute unit will have final study procedures completed at that time and a subsequent office visit will not be required. In all cases, the prescribed rivaroxaban therapy must have been completed prior to the time of the final visit. Safety evaluations at the final visit will include clinical laboratory blood tests, a physical examination, urine pregnancy test (if applicable), recording of any adverse events including details regarding any bleeding episodes or blood clot events, and assessment of the surgical wound. All patients will return any unused study medication and study participation will be complete. All patients will receive oral rivaroxaban 10mg daily. First dose of rivaroxaban will be given within 2 days after admission to the subacute unit, in the morning within 12 hrs (if 30mg twice a day) or 24 hours (if 40mg daily) of the enoxaparin dose. Patients will then continue to receive a daily 10 mg dose each morning. The total duration of combined therapy (enoxparin plus rivaroxaban) may not exceed 35 days for patients with total hip replacement or 14 days with total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* Undergone elective total hip or knee replacement surgery
* Received postoperative venous blood clot prevention therapy within 24 hours of the surgery
* Currently prescribed enoxaparin 30mg subcutaneous (SQ) twice a day or 40mg SQ daily for venous blood clotting prevention with an expected duration of continued prevention therapy of at least 3 days after admission to a subacute unit
* Discharged from the hospital to a subacute unit (including skilled nursing facilities and rehabilitation units) and committed to remaining in the unit for the duration of the Pharmacodynamic blood sampling period of the study

Exclusion Criteria:

* Platelet count <90,000/µL based on screening laboratory assessments
* active internal bleeding or high risk of bleeding
* history of, or condition associated with, increased bleeding risk including
* planned invasive procedure with potential for uncontrolled bleeding, including major surgery
* sustained uncontrolled high blood pressure, defined as systolic blood pressure =180 mmHg or diastolic blood pressure =100 mmHg
* clinically significant kidney disease and/or impaired kidney function
* clinically significant liver disease
* anemia
* known allergies, hypersensitivity, or intolerance to rivaroxaban
* indication for anticoagulant (blood thinning) therapy for a condition other than blood clot prevention
* anticipated need for treatment with a prescription or nonprescription non-steroidal anti-inflammatory drugs (NSAIDs)
* any patient who has taken more than one or two doses of aspirin (>100 mg/dose) in the week prior to enrollment will not be allowed to participate
* Drug addiction or alcohol abuse within 3 years prior to screening

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ortho-McNeil Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Ortho-McNeil Janssen Scientific Affairs, LLC
Locations (5):
- United States (5):
  - Denver, Colorado
  - Hollywood, Florida
  - Tamarac, Florida
  - Vero Beach, Florida
  - Glen Cove, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Rivaroxaban: 10 mg PO (orally) qd (once daily) for up to 35 days for total hip replacement (THR) and 14 days for total knee replacement (TKR)
Period: Overall Study
Arm/Group | Rivaroxaban
Started | 53
Completed | 46
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Groups:
- Rivaroxaban: 10 mg PO qd for up to 35 days for THR and 14 days for TKR
Arm/Group | Rivaroxaban
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (11.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 24
Region of Enrollment [Number; unit: participants]
  UNITED STATES | 53
Surgical Type [Number; unit: participants]
  Hip | 26
  Knee | 27
Baseline BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.5 (6.78)
Baseline Estimated Glomerular Filtration Rate (eGFR) From Local Lab [Number; unit: participants]
  eGFR >= 60 mL/min | 47
  eGFR Between 30 and 59 mL/min | 6
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 52

OUTCOME MEASURES:

1. Primary Outcome: Summary of Change From Day 3 to Day 1 in Maximum Anti-Factor Xa (aFXa)
Description: Descriptive statistics for per-patient maximum Anti-Factor Xa laboratory value selected from the 7 consecutive blood draws (0, 2, 4, 6, 8, 12 and 24 hrs post dose) on Day 1 and Day 3
Time Frame: Day 1, Day 3
Population: ITT population: All subjects who received study drug and had valid post-dose data collected for efficacy analysis.
Measure: Mean (Standard Deviation); unit: IU/ml
Arm/Group | Rivaroxaban
Number analyzed (Participants) | 52
IU/ml
  Day 1 | 1.66 (0.422)
  Day 3 | 1.83 (0.305)
Statistical Analysis 1: Comparison: Rivaroxaban; Test type: Superiority or Other; p = .008, t-test, 2 sided; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [-0.05 to 0.34], Standard Deviation 0.5

2. Primary Outcome: Summary of Change From Day 3 to Day 1 in Maximum Prothrombin Time
Description: Descriptive statistics for per-patient maximum prothrombin time laboratory value selected from the 7 consecutive blood draws (0, 2, 4, 6, 8, 12 and 24 hrs post dose) on Day 1 and Day 3
Time Frame: Day 1, Day 3
Population: ITT population: All subjects who received study drug and had valid post-dose data collected for efficacy analysis
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Rivaroxaban
Number analyzed (Participants) | 52
sec
  Day 1 | 21.57 (3.405)
  Day 3 | 20.51 (3.179)
Statistical Analysis 1: Comparison: Rivaroxaban; Test type: Superiority or Other; p = 0.111, t-test, 2 sided; Mean Difference (Final Values) = -0.91, 95% CI 2-sided [-2.048 to 0.219], Standard Deviation -1.10

3. Secondary Outcome: Summary of Change From Day 1 to Day 3 in Area Under the Curve (AUC) of aFXa
Description: Descriptive statistics for Area Under the Curve (AUC) on Study Day 1 and Day 3 for Anti-Factor Xa, based on the 7 consecutive blood draws at 0, 2, 4, 6, 8, 12 and 24 hours post dose
Time Frame: Day 1, Day 3
Population: ITT population: All subjects who received study drug and had valid post-dose data collected for efficacy analysis
Measure: Mean (Standard Deviation); unit: IU/ml*hour
Arm/Group | Rivaroxaban
Number analyzed (Participants) | 52
IU/ml*hour
  Day 1 | 21.35 (7.086)
  Day 3 | 20.74 (7.17)
Statistical Analysis 1: Comparison: Rivaroxaban; Test type: Superiority or Other; p = 0.87, t-test, 2 sided; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-2.77 to 2.35], Standard Deviation 6.977

4. Secondary Outcome: Summary of Change From Day 1 to Day 3 in AUC of Prothrombin Time
Description: Descriptive statistics for AUC on Study Day 1 and Day 3 for prothrombin time, based on the 7 consecutive blood draws at 0, 2, 4, 6, 8, 12 and 24 hours post dose
Time Frame: Day 1, Day 3
Population: ITT population: All subjects who received study drug and had valid post-dose data collected for efficacy analysis
Measure: Mean (Standard Deviation); unit: sec*hour
Arm/Group | Rivaroxaban
Number analyzed (Participants) | 52
sec*hour
  Day 1 | 420.46 (44.361)
  Day 3 | 391.37 (42.664)
Statistical Analysis 1: Comparison: Rivaroxaban; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -35.13, 95% CI 2-sided [-48.01 to -22.26], Standard Deviation 36.316

ADVERSE EVENTS:
Time Frame: 30 days
Description: From the first dose day to the final evaluation day.
Arm/Group | Rivaroxaban
Serious Adverse Events (participants affected / at risk) | 3/53
Other Adverse Events (participants affected / at risk) | 38/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (N=53)
Arthritis Infective (Infections and infestations) | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1
Anxiety (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rivaroxaban (N=53)
Constipation (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 9
Asthenia (General disorders) | 7
Pyrexia (General disorders) | 7
Oedema (General disorders) | 4
Blood Iron Decreased (Investigations) | 5
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 5
Insomnia (Psychiatric disorders) | 5
Fall (Injury, poisoning and procedural complications) | 3
Transfusion (Surgical and medical procedures) | 3

LIMITATIONS AND CAVEATS:
There were 56 subjects enrolled in the study, but only 53 of them were treated with study medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days